CLINICAL TRIAL: NCT05655845
Title: Bowel Function and Risk Factors for Bowel Dysfunction at Preschool and Early Childhood Age in Children With Hirschsprung Disease
Brief Title: Risk Factors for Bowel Dysfunction at Preschool and Early Childhood Age in Children With Hirschsprung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weibing Tang (Other)
Responsible Party: Sponsor-Investigator, Weibing Tang, Clinical Professor, Nanjing Children's Hospital
Organization: Nanjing Children's Hospital (Other)
Other Study IDs: NanjingCH1129
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Bowel Dysfunction; Hirschsprung Disease; Risk Factor; Incontinence; Constipation
Keywords: Hirschsprung Disease; Bowel function; associated factors
MeSH Terms: conditions — Intestinal Diseases; Hirschsprung Disease; Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysfunction group: Bowel function score(BFS,total 20 points) was approved by Rintala in 1995 and patients with a score < 17 were considered to have bowel dysfunction.
  Interventions: Other: bowel function score(BFS) questionnaire survey
- near-normal group: Bowel function score(BFS,total 20 points) was approved by Rintala in 1995 and patients with a score > 17 were considered to have normal bowel habits.
  Interventions: Other: bowel function score(BFS) questionnaire survey

INTERVENTIONS:
Other: bowel function score(BFS) questionnaire survey — A cross-sectional bowel function score(BFS) questionnaire survey was conducted in patients with HD who underwent PTs between January 2014 and December 2019 at Children's Hospital of Nanjing Medical University.Patients consented to the survey were asked to complete the questionnaire,and were divided into two groups: dysfunction group(BFS<17 ); and normal group (BFS>=17 ). The operative age, birth weight, premature delivery status, operative weight, aganglionic segment, single or stage PT, surgical approach(laparotomy or laparoscopy), post-operative Hirschsprung-associated enterocolitis (HAEC),and immediate complications were recorded and compared between two groups。Both univariate and multivariate regression analysis were used to seek the risk factors of bowel dysfunction after PTs in HD. .

SUMMARY:
Bowel dysfunction has been proven as the most common complication after pull-through(PT) of Hirschsprung disease(HD) ，which may persist to adulthood and lead to social problems.The reason of bowel dysfunction is complicated and the risk factors were not defined.

DETAILED DESCRIPTION:
Hirschsprung disease (HD) is a distinctive congenital disease with the absence of ganglion cells in the distal intestine leads to distal bowel obstruction and defecation disorders. HD is a rare disease, with a reported incidence of 1:5,000, requiring proper surgical treatment for the maintenance of normal or near-normal bowel movement.To date, there is insufficient evidence to recommend a preferred or superior method for the surgical repair, and a pull-through with or without laparoscopy was the most common procedure for correction of HD,which may have faster recovery and less rate of complication compared to other surgical approaches.The short or long-term outcomes of HD have been deeply assessed in the past few years,and bowel dysfunction,consist of soling, incontinence and constipation, had been proven as the most common complication,which may be a ongoing issue and lead to social problems,which should not be ignored. Otherwise,there were many reports proved that poor bowel function in preschool and early childhood may lead to social problems and depression in adolescence or adult.Many factors may lead to bowel dysfunction in HD, including length of aganglionic segement,anastomotic leakage or redo-PT,unsuitable timing of surgery,etc.Thus,the present study was designed to seek the risk factors for bowel dysfunction of HD,which is meaningful to maintain or improve the bowel function in preschool and early childhood.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical dignosis with Hirschsprung disease
2. completed the toilet training

Exclusion Criteria:

1. redo-pull-through,
2. Down syndrome or other co-morbidities that impaired functional outcomes

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HD who underwent PTs between January 2014 and December 2019 at Children's Hospital of Nanjing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
bowel function score | through study completion, an average of 5 year
  Bowel function score(BFS,total 20 points) was approved by Rintala in 1995 and patients with a score > 17 were considered to have normal bowel habits. 7 items were in BFS,including ability to hold back defecation,feels/reports the urge to defecate,frequency of defecation,soiling,accidents,constipation.
Clavien-Dindo classifification of surgical complications | through study completion, an average of 5 year
  Clavien-Dindo is an objective grading system, which is used for grading postoperative complications in a reproduceable manner.It consists of five grades ranging from any deviation from a normal postoperative course (Grade I) to death (Grade V)
Hirschsprung disease associated enterocolitis(HAEC) | through study completion, an average of 5 year
  The guidelines for the diagnosis and management of HAEC were defined by the American Pediatric Surgical Association in 2017. There are three types of HAEC defined by severity: possible HAEC [grade I]; definite HAEC [gradeⅡ]; and severe HAEC [grade Ⅲ].

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Tang, Dr, Study Director — Children's Hospital of Nanjing Medical University
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
All data generated or analyzed during this study are available from the corresponding authors upon reasonable request.

REFERENCES:
- [Derived] Pan S, Li W, Shi C, Tang W, Lu C. Features of defecation dysfunction among patients with Hirschsprung disease in early childhood. BMC Gastroenterol. 2025 Jul 9;25(1):510. doi: 10.1186/s12876-025-04106-4. PMID 40634926